CLINICAL TRIAL: NCT01921543
Title: Electrical Stimulation of the Internal Capsule/Grey Matter and Inferior Thalamic Peduncle for Treatment-refractory Major Depressive Disorder
Brief Title: Deep Brain Stimulation in Treatment Refractory Depression
Acronym: DBSTRD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patient inclusion was very tedious and slower than expected. (7 patients in 5 years)
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: s28650
Record Dates: First submitted 2013-01-08; First posted 2013-08-13 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Major Depressive Disorder
Keywords: Deep Brain Stimulation; Major Depressive Disorder; Psychosurgery; Electrical stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CI/BNST stimulation on (Experimental)
  Interventions: Device: CI/BNST stimulation
- CI/BNST vs stimulation off (Experimental): randomized, double blind, 1 week crossover
  Interventions: Device: CI/BNST stimulation; Device: No stimulation
- ITP stimulation on (Experimental)
  Interventions: Device: ITP Stimulation
- CI/BNST vs ITP vs stimulation off (Experimental): randomized, double blind, two month crossover
  Interventions: Device: ITP Stimulation; Device: CI/BNST stimulation; Device: No stimulation

INTERVENTIONS:
Device: ITP Stimulation — Model 7428 Kinetra® Neurostimulator
  Model 3887 DBSTM Pisces Quad Compact Model 3389 DBSTM Brain Lead
  Model 3387 DBSTM Brain Lead
  Model 7482-51 Extension
  Model 7482-66 Extension
  Model 7482-95 Extension
  Model 7436 AccessTM Therapy Controller
  Model 3628 Dual Screener TM
  Model 8840 N'Vision
  Arms: CI/BNST vs ITP vs stimulation off; ITP stimulation on
Device: CI/BNST stimulation — Model 7428 Kinetra® Neurostimulator
  Model 3887 DBSTM Pisces Quad Compact Model 3389 DBSTM Brain Lead
  Model 3387 DBSTM Brain Lead
  Model 7482-51 Extension
  Model 7482-66 Extension
  Model 7482-95 Extension
  Model 7436 AccessTM Therapy Controller
  Model 3628 Dual Screener TM
  Model 8840 N'Vision
  Arms: CI/BNST stimulation on; CI/BNST vs ITP vs stimulation off; CI/BNST vs stimulation off
Device: No stimulation
  Arms: CI/BNST vs ITP vs stimulation off; CI/BNST vs stimulation off

SUMMARY:
The main aim of this trial was to investigate whether patients suffering from treatment refractory- Major Depressive Disorder (MDD) can benefit from DBS (Deep Brain Stimulation) in the brain areas known as inferior thalamic peduncle (ITP) and/or Capsula Interna/Bed nucleus of the stria terminalis (CI/BNST)

DETAILED DESCRIPTION:
This study aims to investigate the effect of deep brain stimulation (DBS)in major depressive disorder (MDD). After implantation of the DBS system, the effects of deep brain stimulation in ITP and CI/BNST will be evaluated.

The design of the study consists of two consecutive crossover phases, interspaced with 2 optimalisation episodes. After a period of optimalisation of CI/BNST stimulation parameters, patients will be randomised in two groups. Half of the group of patients will receive stimulation in CI/BNST. The other half will not. After one week both groups will switch conditions during a period of one week. This will give an idea of the effects of stimulation in CI/BNST on the outcome measures. Outcome measures will be evaluated after each week.

After this first crossover patients will continue to an optimalisation phase of ITP stimulation parameters. A second crossover will then follow. The effects of ITP stimulation, CI/BNST stimulation and no stimulation will be compared. In this phase patients will again be randomised to receive one of the six possible combinations of three consecutive periods of two months for the three different stimulation conditions (ITP stimulation, CI/BNST stimulation and no stimulation).

Evaluations of outcome measures will be performed by blinded evaluators. This design will limit the duration of periods in which these severly ill patients are not stimulated.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder, severe, unipolar type, diagnosed by Structured Clinical Interview for DSM-IV (SCID-IV), judged to be of disabling severity.
* 17-item Hamilton Depression Rating Scale (HDRS) score of at least 19.
* Global Assessment of Function (GAF) score of 45 or less.
* A recurrent (>4 episodes) or chronic (episode duration >2 years) course and a minimum of 5 years since the onset of the first depressive episode. Major impairment in functioning or potentially severe medical outcomes (repeated hospitalizations, serious suicidal ideation or a history of previous suicide attempts or other self-injurious behavior).
* Failure to respond to:

  * adequate trials (>6 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes AND;
  * adequate trials (>4 weeks at the usually recommended or maximum tolerated dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant) AND;
  * an adequate trial of Electroconvulsiontherapy (ECT) (>6 bilateral treatments) AND;
  * adequate relapse prevention by antidepressant medication or maintenance ECT or an adequate trial of individual psychotherapy.
* Age ≥18 - ≤65 years.
* Able to comply with the operational and administrative requirements of participation in the study ; able to comply with the questionnaires and the protocol.
* Able to give written informed consent.
* Either drug-free or on a stable drug regimen for at least 6 weeks at the time of entry into the study.
* Good general health.
* Candidates may have undertaken additional trials of potentially beneficial novel combinations of medication and psychotherapy, or they may have undertaken trials of novel interventions lacking definitive evidence of efficacy in severe depression (e.g., light therapy, herbal therapy, transcranial magnetic stimulation, vagal nerve stimulation).

Exclusion Criteria:

* Current or past non-affective psychotic disorder.
* Any current clinically significant neurological disorder or medical illness affecting brain function.
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
* Any surgical contraindications to undergoing DBS, including labeled contraindications for DBS and/or inability to undergo presurgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation or significant cardiac or other medical risk factors for surgery.
* Current or unstably remitted substance abuse.
* Pregnancy and women of childbearing age not using effective contraception.
* History of severe personality disorder, especially cluster B.
* Imminent risk of suicide (based on the judgment of the investigators)
* Present participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms as measured by the 17-item Hamilton Depression Rating Scale | up to 14 months
  The time frame is an approximation as evaluation is performed after each crossover phase. The time interval between baseline and evaluation depends on the time required for optimisation of DBS parameters.

SECONDARY OUTCOMES:
Montgomery- Asberg Depression Rating Scale (MADRS) | up to 14 months
Inventory for Depressive Symptoms, Self-Report (IDS-SR) | up to 14 months
Global measures of illness severity and improvement:the clinician-rated Clinical Global Impressions - Severity (CGI-S) and Clinical Global Impressions - Improvement (CGI-I) scales, and the patient-rated Patient Global Impressions (PGI-S and PGI-I) | up to 14 months
Global Assessment of Function (GAF) | up to 14 months
patient-rated Symptom CheckList (SCL-90) | up to 14 months
Cognitive function: Rey Auditory Verbal Learning Test; Trailmaking A & B, Stroop Test, Rey-Osterrieth complex figure test ; Wisconsin Card Sorting Test; Standard Progressive Matrices of Raven; Digit Span Test; Word Fluency Test | up to 14 months
Hopelessness: using the Beck Hopelessness scale | up to 14 months
Hamilton Anxiety Rating Scale (HARS) | up to 14 months
Young Mania Rating Scale (YMRS) | up to 14 months
Side Effects Questionnaire (SEQ) | up to 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium